CLINICAL TRIAL: NCT04312308
Title: A Study for Identification of Predictive Immune Biomarker for Atezolizumab Therapy in NSCLC Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Other Study IDs: 4-2019-0948
Record Dates: First submitted 2020-02-28; First posted 2020-03-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Immune biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Small Cell Lung Cancer Treated with Atezolizumab: Patients with Non-Small Cell Lung Cancer Treated with Atezolizumab
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — 1. .Analysis of immune marker using FACS before treatment and Cycle1, Cycle2, Cycle3 and the time of disease progression.
  2. .Multiplexed biomarker analysis of tumor and immune cells in tumor microenvironment (TME) at pre-treatment and progression (Pre-treatment biopsy is mandatory but biopsy is optional for disease progression)
  3. microbiome Pretreatment stool sample will be collected. (Stool sample is optional)
  4.Genetic analysis For RNAseq or exome seq, biopsied tissue at baseline or progression are optional.
  4.Single cell RNA sequencing (scRNA-seq) scRNA-seq will be performed by collecting selectively tissues from pre-treatment tumor biopsies and at relapse/acquired resistance tumor biopsies. Screening and treatment biopsies are optional.

SUMMARY:
The study aimed to elucidate predictive immune related biomarker to the responsiveness to the PD-L1 blockade and evaluate the dynamics of immune cells in peripheral blood from NSCLC patients during atezolizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   a) Subjects must have signed and dated an IRB/IEC-approved written informed consent form in accordance with regulatory and institutional guidelines.
2. Target Population

   1. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1
   2. Subjects with histologically- or cytologically-documented NSCLC who presented with Stage IIIB/Stage IV disease and who have relapsed after treatment for stage IIIB/stage IV disease following chemotherapy, radiation therapy, or surgical resection.
   3. Subjects must have disease progression or recurrence during or after at least 1 systemic therapy for advanced or metastatic disease.

   i) Each subsequent line of therapy must be preceded by disease progression. ii) Subjects who received platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, and developed recurrent (local or metastatic) disease within 6 months of completing therapy are eligible.

   iii) Subjects with recurrent disease > 6 months after completing a platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, who also subsequently progressed during or after a systemic regimen given to treat the recurrence, are eligible.

   d) Prior chemotherapy or TKI therapy must have been completed at least 1 week before study drug administration. All AEs due to prior chemotherapy or immunotherapy have either returned to baseline or stabilized.

   e) Prior palliative radiotherapy must have been completed at least 7 days prior to study drug administration.

   f) Subjects are eligible if CNS metastases are treated or subjects have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 14 days prior to enrollment. In addition, subjects must either be off corticosteroids or on a stable dose or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) g) Screening laboratory values must meet the following criteria prior to commencement of treatment: i) WBCs ≥ 2000/µL ii) Neutrophils ≥1500/µL iii) Platelets ≥ 100 X10³/µL iv) Hemoglobin ≥ 9.0 g/dL v) Serum creatinine of ≤ 1.5 X ULN or creatinine clearance (CrCl) > 40 mL/minute (using Cockcroft/Gault formula)

(1). Female CrCl= [(140- age in years) X weight in kg X 0.85) ÷ (72 X serum creatinine in mg/ dL)] (2). Male CrCl= [(140- age in years) X weight in kg X 1.00) ÷ (72 X serum creatinine in mg/ dL)] vi) AST and ALT ≤ 3 X ULN (In the case of patients with liver metastasis, AST (GOT) and ALT (GPT) ≤ 5.0 times the upper limit of normal range) vii) Total bilirubin ≤ 1.5 X ULN (except subjects with Gilbert Syndrome, who must have total bilirubin < 3.0 mg/dL) h) Subjects with Type I diabetes mellitus, residual hypothyroidism due to an autoimmune condition requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

i) Subjects with available PD-L1 immunohistochemistry (IHC) result could be enrolled regardless of the results of PD-L1 IHC.

j) Subject re-enrollment: This study permits the re-enrollment of a subject who has discontinued the study as a pre-treatment failure (ie, subject has not been treated). If re- enrolled, the subject must be re-consented.

3. Age and Reproductive Status

1. Men and women aged ≥ 18 years old
2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
3. Women must not be breastfeeding
4. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with atezolizumab plus 5 half-lives of atezolizumab (5 x half-life = 135 days) plus 30 days (duration of ovulatory cycle) for a total of 165 days or 24 weeks post-treatment completion.
5. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with atezolizumab plus 5 half-lives of the study drug (135 days) plus 90 days (duration of sperm turnover) for a total of 32 weeks post-treatment completion.
6. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, subjects must agree to the use of 2 methods of contraception, with 1 method being highly effective and the other method being either highly effective or less effective as listed below:

HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

* Male condoms with spermicide
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by WOCBP subject or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug.
* Non-hormonal IUDs, such as ParaGard®
* Tubal ligation
* Vasectomy
* Complete abstinence NOTE: Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs.

Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternative methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

LESS EFFECTIVE METHODS OF CONTRACEPTION

* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal sponge
* Male condom without spermicide
* Progestin only pills by WOCBP subject or male subject's WOCBP partner
* Female condom
* NOTE: A male and female condom must not be used together

Exclusion Criteria:

a) Target Disease Exceptions i) Subjects with ECOG PS ≥ 2 ii) Subjects with untreated CNS metastases are excluded. Subjects are eligible if CNS metastases are treated or subjects have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. In addition, subjects must either be off corticosteroids or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).

iii) Subjects with carcinomatous meningitis are excluded iv) Subjects with < 6 weeks life expectancy b) Medical History and Concurrent Diseases i) Subjects with known active, known, or suspected autoimmune disease which the investigator considers significant ii) Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first dose of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.

iii) Subjects who received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CT137 or anti-CTLA-4 antibody including ipilimumab or any other antibody or drug specifically targeting T cell costimulation or checkpoint pathways iv) Subjects with interstitial lung disease. v) Other active malignancy requiring concurrent intervention vi) Subjects with previous malignancies (except non-melanoma skin cancers and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 1 year prior to study entry AND no additional therapy is required during the study period vii) Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive protocol therapy viii) All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 5) or baseline before administration of study drug ix) Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment x) Known alcohol or drug abuse

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-Small Cell Lung Cancer Treated with Atezolizumab
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
To explore early biomarker to predict response and overall survival after Atezolizumab therapy | up to 1year
  Analysis of immune marker using FACS
To explore early biomarker to predict response and overall survival after Atezolizumab therapy | up to 1year
  Multiplexed biomarker analysis of tumor and immune cells in tumor microenvironment (TME) (Pre-treatment biopsy is mandatory but biopsy is optional for disease progression)
To explore early biomarker to predict response and overall survival after Atezolizumab therapy | up to 1year
  microbiome
To explore early biomarker to predict response and overall survival after Atezolizumab therapy | up to 1year
  Genetic analysis
To explore early biomarker to predict response and overall survival after Atezolizumab therapy | up to 1year
  Single cell RNA sequencing (scRNA-seq)

SECONDARY OUTCOMES:
ORR(Objective response rate) | Atezolizumab treatment will be given every 3 weeks up to progression or 1 year. The manner and interval of efficacy assessment for tumor scan will depends on the investigator's decision.
  The manner and interval of efficacy assessment for tumor scan will depends on the investigator's decision.
PFS(Progression free survival) | Atezolizumab treatment will be given every 3 weeks up to progression or 1 year. The manner and interval of efficacy assessment for tumor scan will depends on the investigator's decision.
  The manner and interval of efficacy assessment for tumor scan will depends on the investigator's decision.
OS(Overall survival) | Overall survival will be followed continuously while subjects are on the study drug and every 6 months after discontinuation or progression for up to 5 years
  Overall survival will be followed continuously while subjects are on the study drug and every 6 months after discontinuation or progression for up to 5 years following the start of therapy either by direct contact (office visits) or via telephone contact, until death, withdrawal of study consent, or lost to follow-up. Overall survival is defined as the time between the start of treatment and the date of death due to any cause.
Safety | local laboratory assessments should be done with prior to each atezolizumab dose Atezolizumab treatment will be given every 3 weeks up to progression or 1 year.
  Number of participants with adverse events and abnormal laboratory values as assessed by NCI-CTCAE version 5

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided